CLINICAL TRIAL: NCT05080244
Title: Evaluation of the Efficacy of Probiotics Taken During the Acute Phase of COVID-19 to Reduce the Occurrence of Long COVID
Brief Title: WHO COVID-19 - Evaluation of the Efficacy of Probiotics to Reduce the Occurrence of Long COVID
Acronym: PROVID-LD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-3700-ECR
Record Dates: First submitted 2021-09-28; First posted 2021-10-15 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: Long COVID; COVID-19; Sars-CoV-2; Coronavirus; Probiotics
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Coronavirus Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Two probiotic strains will constitute the experimental arm (Probiotics). Participants will take two capsules per day (one closed capsule to swallow and one open capsule mixed with maple syrup) for 10 days and one closed capsule per day to swallow for the following 15 days. They will stop the treatment if they are admitted to the hospital. The treatment will last a maximum of 25 days.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Potato starch and magnesium stearate will constitute the comparator arm (Placebo). Participants will take two capsules per day (one closed capsule to swallow and one open capsule mixed with maple syrup) for 10 days and one closed capsule per day to swallow for the following 15 days. They will stop the treatment if they are admitted to the hospital. The treatment will last a maximum of 25 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — 2 strains 10x10^9 UFC/capsule
  Arms: Probiotics
Dietary Supplement: Placebo — Potato starch and magnesium stearate
  Arms: Placebo

SUMMARY:
Probiotics may be considered as an option of treatment for long COVID since they have anti-viral effect, trigger immunomodulation and have low side-effects. This randomized controlled trial aims to reduce the number of patients with long COVID by 25% 90 days after the COVID-19 diagnosis by taking probiotics in a symptomatic population, self-caring at home. During the acute phase of the disease, participants will take two capsules (probiotics or placebo) per day for 10 days and one capsule (probiotics or placebo) per day for the following 15 days. A follow-up will be done twice during the acute phase, 14 days and 28 days after starting to take the investigational product (compliance to treatment, side effects, etc.). At inclusion and at Day14, Day30 and Day90 after the COVID-19 diagnosis, a questionnaire will be administered (COVID-19 symptoms, anxiety, functioning difficulties, etc.) and 2 saliva and 2 stool (viral and microbiota analyzes) self-samples will be performed.

DETAILED DESCRIPTION:
Rational:

COVID-19 disease caused by a new coronavirus (SARS-CoV-2) has received worldwide attention. No effective treatment against COVID-19 is available and the current vaccination appears essential to control the pandemic. However, many questions remain, such as the durability of immunity and the appearance of variants. While the acute phase has been widely studied, the long-term consequences are unknown, and a new burden is emerging: the long COVID. The long COVID is defined by the persistence of symptoms of the disease for more than 4 weeks after diagnosis. Several strong arguments support the study of probiotics for COVID-19: 1) probiotics act on viruses by various well described mechanisms (reduction of absorption, cellular internalization of the virus, production of metabolites/substances having a direct antiviral effect and immunomodulation); 2) probiotics are considered with a high level of evidence (meta-analysis) to reduce diarrhea (associated with antibiotics and Clostridium difficile) and for respiratory tract infections and 3) probiotics are affordable and available with low side-effects.

Objectives:

Primary objective: Reduce by 25% the number of patients with LONG-COV during follow-up at D90 by taking probiotics during the acute phase of COVID-19.

Secondary objectives (Obj S):

Objective S1: Compare the proportion of patients presenting COVID-19 symptoms and severity of symptoms at D14, D30 and D90 by taking probiotics during the acute phase of COVID-19.

Objective S2: Describe the symptoms severity and evolution by study group and baseline characteristics.

Objective S3: Determine/identify prognostic factors measured at baseline (inclusion) associated with LONG-COV (sociodemographic, clinical factors).

Population:

618 men and women, 18 years or older, with a first positive test for COVID-19 in the last 10 days, having symptoms of the COVID-19, self-caring at home, living in Quebec for the next 90 days, able to take medication alone, with access to a phone or to the Internet.

Randomization:

Patients will be randomized in one of the study groups (stratified by age and gender). The randomization is double-blinded and uses a ratio 1:1. Group A: will take probiotics for 25 days / Group B: will take placebo for 25 days.

Intervention:

During the acute phase of the disease, participants will take two capsules (probiotics or placebo) per day (one closed capsule to swallow and one open capsule mixed with maple syrup) for 10 days and one closed capsule (probiotics or placebo) per day to swallow for the following 15 days.

Data collection:

A follow-up will be done twice during the acute phase, 14 days and 28 days after starting to take the investigational product to evaluate compliance to treatment, medication intake, side effects, etc. At inclusion and at Day14, Day30 and Day90 after the COVID-19 diagnosis, the participant will complete a questionnaire that will focus on COVID-19 symptoms, food intake, anxiety, functioning difficulties, quality of life, etc. For those who will be admitted to hospital, data on their admission, complications and treatments will be collected.

Definition of LONG-COV:

The status of FLU-PRO and quality of life indicators before COVID-19 disease was initially unknown. Thus, we have operationalized the WHO's definition to select patients. If at least one of the criteria was met (see SAP for details), the participant would be qualified for an expert's review.

Every diagnosis based on Binomes was reviewed by expert on LONG-COV physicians. Those initially selected who potentially qualified for LONG-COV were called after the study to verify if symptoms were present or not before the positive detection of COVID-19. The final decision was on the expert physician responsibility.

Samples:

At inclusion and at Day14, Day30 and Day90 after the COVID-19 diagnosis, 2 saliva and 2 stool (viral and microbiota analyzes) self-samples will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* ≤ 10 days between the COVID-19 diagnosis and the inclusion
* Having symptoms of the COVID-19 at inclusion
* Living in Quebec for the next 90 days
* Self-caring at home
* Able to take medication alone
* With access to a phone or to the Internet
* Able to give informed consent

Exclusion Criteria:

* Taking probiotic supplements at inclusion
* Taking antibiotics for a reason other than COVID-19 at inclusion
* Allergies to soy, lactose, yeast, maltodextrin, vitamin C, potato starch, magnesium stearate, hypromellose or titanium dioxide
* Has a chronically weakened immune system (AIDS, lymphoma, chemo-radio-corticosteroid therapy, immunosuppressive pathology)
* Was treated with chemo-radio-corticosteroid therapy in the last 6 months
* Has active cancer
* Taking immunosuppressive drugs (e.g. anti-rejection treatment after organ transplant)
* Already participating in another randomized clinical trial
* Is pregnant, expects to become pregnant in the next few months or is breastfeeding
* Has any other condition that would prevent safe participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Reduce by 25% the number of patients with LONG-COV during follow-up at D90 by taking probiotics during the acute phase of COVID-19 | 90 days after the COVID-19 diagnosis.
  COVID-19 symptoms (FLU-PRO), anxiety (GAD-7) and functioning difficulties (WG-SS)

SECONDARY OUTCOMES:
Compare the proportion of patients presenting COVID-19 symptoms and severity of symptoms at D14, D30 and D90 by taking probiotics during the acute phase of COVID-19. | 14,30 and 90 days after the COVID-19 diagnosis.
  COVID-19 symptoms (FLU-PRO), anxiety (GAD-7) and functioning difficulties (WG-SS)
Describe the symptoms severity and evolution by study group and baseline characteristics. | Inclusion, Day14, Day30 and Day90 after the COVID-19 diagnosis
  COVID-19 symptoms (FLU-PRO), baseline characteristics
Determine/identify prognostic factors measured at baseline (inclusion) associated with LONG-COV (sociodemographic, clinical factors). | Inclusion, Day14, Day30 and Day90 after the COVID-19 diagnosis
  COVID-19 symptoms (FLU-PRO), anxiety (GAD-7) and functioning difficulties (WG-SS), baseline characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — CIUSSSE-CHUS
Locations (1):
- CIUSSS de L'Estrie-CHUS Hospital, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT05080244/SAP_001.pdf